CLINICAL TRIAL: NCT07194993
Title: Defining Protein Requirements in Adults With PKU: Impact of Genotype and Medical Food Intake
Brief Title: PKU Protein Requirements
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Rani Singh, Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00009869
Record Dates: First submitted 2025-09-19; First posted 2025-09-26 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: PKU

STUDY DESIGN:
Intervention Model Description: The Primary purpose of this study is focused on Translational Science. The study will determine the protein requirements in one group of participants with PKU, based on genotype and medical food consumption, using the IAAO method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Adults with PKU receiving test diet and Oral stable nonradioactive isotope provision (Experimental): Participants will receive amino acid tracer (Oral stable nonradioactive isotope provision) and test diet (medical food) throughout each study day, for a total of 7 study days.
  Interventions: Other: Nonradioactive stable oral isotope; Other: Test diet

INTERVENTIONS:
Other: Nonradioactive stable oral isotope — NaH13CO3 [99% atom percent excess (APE) and L-[1-13C]Leu (99% APE) will be given orally.
  Isotope administration will begin with the fifth meal on each study day with each remaining meal.
  The nonradioactive stable oral isotope is being administered to study the physiological process of amino acid oxidation.
  Other Names: Oral Isotope tracer
Other: Test diet — Test diets will be provided on study days in 8 hourly isocaloric and isonitrogenous meals to maintain a metabolic steady state.
  Each meal will provide one-twelfth of the participant's daily needs to model a 12-hour fasted and 12-hour fed feeding pattern.
  The diet will be composed of PFD2 (Mead Johnson), Tang and Kool-Aid (Kraft), corn oil, and protein-free wheat starch cookies. Each participant will receive 1 of 7 test protein intakes (0.2-3.2 g ⋅ kg-1 ⋅ d-1) on each study day. Protein will be provided as a crystalline L-amino acid mixture based on an egg protein pattern. Phe will be provided separately based on the Phe tolerance for each patient established by the metabolic dietitian listed on the IRB protocol. Leucine will be provided at a constant amount of 82.6 mg/kg/day as it is used as the indicator amino acid. The medical food used in this study is being fed to subjects for nutritional purposes to study the oxidation of the nonradioactive oral isotope.
  Other Names: Medical Food

SUMMARY:
The objective of this research is to determine the protein requirements based on genotype and medical food consumption in a sample of adults with Phenylketonuria (PKU) using the indicator amino acid oxidation (IAAO) method.

DETAILED DESCRIPTION:
Current phenylketonuria (PKU) protein guidelines are based on outdated methods and do not account for differences in genetics or how much medical formula an individual consumes. This research aims to determine more accurate and personalized protein requirements in adults with PKU that have different genetic changes using a safe and direct method called the indicator amino acid oxidation technique. The study will address two specific aims: Aim 1 will determine the protein requirements of adults with PKU that have different genetic changes and Aim 2 will investigate how the ratio of medical formula to protein intake from natural foods affects protein needs.

Adults with PKU will be recruited for this study, and vulnerable populations will not be included.

This study includes surveys, anthropometric measurements, body composition analysis, indirect calorimetry, diet history, collection of blood, urine, and expired breath samples, administration of study day diets and an oral stable isotope protocol.

Recruitment will be at Emory Genetics Clinic. Informed consent will be obtained with an in-person signature or by an electronic IRB approved signature. Participants will attend one preliminary visit and 7 study days. Each study day will last 8 hours. Participants will be enrolled for approximately 4-6 months.

Participants will have the option to bank plasma and urine samples for future use.

ELIGIBILITY:
Inclusion Criteria:

* will be males and females (50:50) 18 years and older who were diagnosed with PKU through newborn screening or diagnosis later in life, capable of providing consent, and have previously had mutation testing

Exclusion Criteria:

* include concurrent illness, recent history of weight loss or acute illness during the past 6 months that could affect protein metabolism, pregnancy, lack of regular menstruation, implantable electronic devices or pacemakers, history of claustrophobia, and inability to provide consent. In addition, participants will be excluded if their genotype subgroup has already reached its predefined maximum enrollment (n=4)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Change in rate of oxidation of tracer in the expired breath | Baseline, post-intervention (3-8 hours post-baseline)
  The rate of oxidation of tracer in the expired breath will be measured in each study day.

SECONDARY OUTCOMES:
Change in Phenylalanine concentrations before and after provision of the oral isotope protocol to provide an assessment of phenylalanine and tyrosine metabolism following study day | Baseline, post-intervention (8 hours post-baseline)
  Phenylalanine concentration before and after provision of the oral isotope protocol to provide an assessment of phenylalanine metabolism following study day diets.
Change in Tyrosine concentrations before and after provision of the oral isotope | Baseline, post-intervention (8 hours post-baseline)
  Tyrosine concentrations before and after provision of the oral isotope protocol to provide an assessment of tyrosine metabolism following study day diets.
Ratio of medical food protein to protein from foods protein to protein from foods | Throughout the study (Up to 6 months post-intervention)
  Ratio of medical food protein to protein from foods as reflected on 3-day diet records throughout the study.
Number of participants with no adverse events related to study day diets and nonradioactive isotope tracers | End of study (Up to 6 months post-intervention)
  Tolerability of the study day diet and the oral isotope tracer, primarily gastrointestinal tolerability will be obtained by recording the number of participants with absence of adverse events related to study day diets or nonradioactive isotope tracers.

CONTACTS AND LOCATIONS:
Overall Officials: Rani Singh, PhD, RDN, LD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No